CLINICAL TRIAL: NCT03792997
Title: A Therapeutic Protocol in Previous Failed ART Patients With High Total NK Cells: A Randomized Controlled Trial
Brief Title: A Therapeutic Protocol in Previous Failed ART Patients With High Total NK Cells
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Benha University (Other)
Collaborators: Hawaa Fertility Center (Other)
Responsible Party: Principal Investigator, Ahmed Saad, Assistant professor of Ob. & Gyn., Benha University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Hawaa-6
Record Dates: First submitted 2019-01-02; First posted 2019-01-04 (Actual); Last update posted 2022-01-03 (Actual); Status verified 2021-12

CONDITIONS: Unexplained Infertility
MeSH Terms: interventions — Combined Modality Therapy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- control (Active Comparator): regular treatment with embryo transfer in the form of progesterone I.M. & Supp. in addition to low dose aspirin & folic acid
  Interventions: Combination Product: combination therapy for high peripheral NK cells
- study (Experimental): regular treatment with embryo transfer in the form of progesterone I.M. & Supp. in addition to low dose aspirin & folic acid but the investigators add in this arm lipid emulsion & prednisolone & LMWH
  Interventions: Combination Product: combination therapy for high peripheral NK cells

INTERVENTIONS:
Combination Product: combination therapy for high peripheral NK cells — lipid emulsion & prednisolone & LMWH

SUMMARY:
patients with previous failed ART cycles with high peripheral NK cells will be divided into 2 groups: one group of patients with previous failed ART cyles will undergo standard treatment but the other group will have in addition lipid emulsion &prednisolone & LMWH

DETAILED DESCRIPTION:
patients with previous failed ART cycles with high peripheral NK cells will be divided into 2 groups: one group of patients with previous failed ART cyles will undergo standard treatment but the other group will have in addition lipid emulsion begin in the cycle before embryo transfer &prednisolone begin with the start of lipid emulsion & LMWH begin with the day of ET

ELIGIBILITY:
Inclusion Criteria:

* patients with high peripheral NK cells > 10% unexplained infertility cases cases with endometriosis

Exclusion Criteria:

* uterine factors poor responders< 3 MII oocytes severe male factor & Azospermia

Ages: 20 Years to 37 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — Infertile females undergoing ART cycles
Enrollment: 100 (Actual)
Dates: Start 2019-01-01 (Actual); Primary Completion 2019-12-15 (Actual); Study Completion 2021-12-10 (Actual)

PRIMARY OUTCOMES:
chemical pregnancy rate | 14 days
  quantitative serum test

SECONDARY OUTCOMES:
clinical pregnancy rate | 6 weeks of pregnancy
  gestational sac and fetal echo by ultrasound

CONTACTS AND LOCATIONS:
Overall Officials: ahmed sa saad, MD, ph D, Principal Investigator — Hawaa Fertility Center
Locations (1):
- Banha University- Hawaa Fertility center, Banhā, Qalyubia Governorate, Egypt

IPD SHARING:
Plan to Share IPD: Yes
study protocol, statistical analysis & results
Supporting Information: Study Protocol, CSR
Time Frame: 1 month after publication, for 6 months
Access Criteria: for researchers doing metanalysis.by contacting us by email